CLINICAL TRIAL: NCT06994117
Title: Expanded Access for Mezigdomide
Status: Available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA057-1024; CA057-1070 (Other: BMS Protocol ID)
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Mezigdomide — Mezigdomide
  Other Names: BMS-986348; CC-92480

SUMMARY:
This is an expanded access designed to provide access to Mezigdomide for eligible participants.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: EAP Investigator Requests — http://www.bms.com/clinical_trials/investigator_sponsored_research/Pages/expanded-access-program.aspx